CLINICAL TRIAL: NCT01043614
Title: Project PEER: Peer Education, Exercising and Eating Right
Brief Title: Peer Education, Exercising and Eating Right - Obesity Prevention in Freshmen Women
Acronym: ProjectPEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Ellen M. Evans, Ph.D., Associate Professor, Principal Investigator, University of Illinois at Champaign-Urbana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-04574
Record Dates: First submitted 2009-12-10; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: Obesity; Obesity Prevention; Freshman women; Freshman 15 weight gain; Self efficacy; Activity and nutrition intervention; Peer education
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peer group education (Experimental): Small groups of female college freshmen facilitated by peer educators
  Interventions: Behavioral: PEER group intervention

INTERVENTIONS:
Behavioral: PEER group intervention — An exercise and nutrition intervention that is based on self-efficacy principles and delivered primarily by peer educators to reduce the risk for obesity in female college freshman over one academic year

SUMMARY:
Project PEER utilizes a randomized controlled study design to investigate the combined effects of an exercise and nutrition intervention that is based on self-efficacy principles and delivered primarily by peer educators to reduce the risk for obesity in female college freshman over one academic year (N = 300). The control group will receive minimal interaction from the research team, paralleling the typical freshman experience on the UIUC campus. Recruitment will take place in two waves (consecutive fall terms with n = 150).

During the final year (Fall 2010) of the project, a General Education course will be offered that targets weight management. Importantly, the discussion groups for this course will be taught by peer educators trained using the peer resources further refined during the PEER project. In addition to conventional measures of content knowledge assessed in the college classroom when obtaining class credit, personal physical activity and nutrition behaviors along with behavioral determinants (self-efficacy, self-regulatory skills and outcome expectations) will also be assessed.

Primary Aim 1: To determine the effectiveness of a peer-delivered self efficacy-based behavioral intervention to enhance nutrition and physical activity behaviors and subsequently weight management success in female university freshman over one academic year. We hypothesize that freshmen randomized to the intervention group will be more successful in losing or maintaining weight than the control group through a combination of diet and physical activity strategies.

Primary Aim 2: To examine the role played by social cognitive factors in changing nutrition and physical activity behaviors across one academic year. We hypothesize that self-efficacy will have both a direct influence on behavior and an indirect effect through its influence on self-regulatory skills and outcome expectations.

ELIGIBILITY:
Inclusion Criteria:

* Female
* In first year on campus, enrolled full-time, and in residence on the UIUC campus
* Aged 17-19 yrs (minors will be required to obtain parental signature on the IRB form)
* Free from any chronic disease/condition that would alter ability to exercise or preclude diet manipulation such as diabetes, hypertension or pregnancy.
* Free from an eating disorder as assessed using the Eating Disorder Inventory
* Free from any medications that would alter adiposity or psychological outcomes
* Sedentary or participation in non-professional recreational activity
* Non-smoking
* Body mass index (BMI) between the 50th and 95th BMI-for-age percentile

Exclusion Criteria:

* Male
* Status other than freshman or enrolled for entire year
* Not living on campus
* Smoking
* Pregnant
* Competitive athlete
* Chronic condition that would alter ability to exercise or preclude diet manipulation such as diabetes, hypertension
* Eating disorder as assessed using the Eating Disorder Inventory
* Taking medications that would alter adiposity or psychological outcomes
* Participation in competitive athletics
* BMI outside parameters

Ages: 17 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measures (eg; weight, hip/ waist dimensions) | Baseline, 3 mo, 8 mo, 1 y and 2 y follow up

SECONDARY OUTCOMES:
Self-efficacy measures for physical activity, nutrition | Baseline, 3 mo, 8 mo, 1 y and 2 y follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Evans, PhD, Principal Investigator — Uiversity of Illinois at Urbana- Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States